CLINICAL TRIAL: NCT06539494
Title: Luminal Fructose Kinetics (MARTINI) (2024)
Brief Title: Luminal Fructose Kinetics (MARTINI Study)
Acronym: MARTINI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Max Nieuwdorp, Principle Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL85966.018.23
Record Dates: First submitted 2024-07-18; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: MASLD
Keywords: Fructose; MASLD; Ethanol
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: 2x 11 participants will be given the same intervention (omeprazol daily)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteer (Active Comparator): healthy volunteers who will get omeprazol daily 2dd40 mg for 4 weeks
  Interventions: Drug: Omeprazole 40 MG
- Sujbects with MASLD (Active Comparator): Patients with MASLD who will get omeprazol daily 2dd40 mg for 4 weeks
  Interventions: Drug: Omeprazole 40 MG

INTERVENTIONS:
Drug: Omeprazole 40 MG — Proton pump inhibitor twice a day for 4 weeks

SUMMARY:
In this study the investigators aim is to explore the dynamics of (small) intestinal fructose catabolism in humans and ethanol production in relation to small intestinal signalling pathways and changes in pH, using 13C fructose isotope tracing techniques complemented with direct luminal sampling via small intestinal catheter in biopsy proven MASLD/MASH patients vs healthy (BMI<25) subjects. Additionally the investigators will repeat the experiment after four weeks of administering omeprazole at a dose of 40 mg twice daily. Omeprazole is a proton pump inhibitor, known to elevate pH from 2-6.

DETAILED DESCRIPTION:
The investigators will perform a non blinded single centre intervention study in 2x 11 participants

Participants will be either healthy volunteers with a BMI < 25 and Age 18-65 or patients with MASLD with a BMI >25, Age 18-65

The objective of the investigators is to study the fructose host/microbial kinetics in humans and to establish the role of (small) intestinal pH on fructose fermentation and endogenous ethanol production in a MASLD/MASH population versus healthy subjects

Subjects will be given omeprazole orally given twice a day 40mg for four weeks

At baseline and after four weeks of omeprazole, a fructose challenge test with labelled fructose and fomepizole and a gastroscopy will be performed, during which a nasal-intestinal catheter will be placed to allow for luminal sampling during the fructose challenge test.

ELIGIBILITY:
Inclusion Criteria:

In case of the healthy subject group:

* Adult individuals, age > 18 <65 years
* Male or postmenopauzal females
* BMI <25
* Ability to give informed consent In case of the MASLD/MASH group
* Adult individuals, age > 18 <65 years
* Male or postmenopauzal females
* BMI > 25
* Biopsy proven MASLD/MASH
* Ability to give informed consent

Exclusion Criteria:

* History of sustained excess alcohol ingestion: daily consumption >30g/day (3 drinks per day) for males and >20 g/day (2 drinks per day) for females
* Patients with diabetes
* Bariatric surgery
* Other forms of liver disease (e.g. Hepatitis B,C, Wilson disease, hemochromatosis)
* Proton-pump inhibitor usage one year prior to study participation
* GLP1, SGLT2i or insulin use
* Antibiotic use for the past 3 months
* Probiotic or symbiotic usage
* Pregnant women
* Chronic illness (including a known history of heart failure, renal failure (eGFR <30 ml/min), pulmonary disease, gastrointestinal disorders, or hematologic diseases), or other inflammatory diseases
* Active infection
* Use of ascal, clopidogrel or other platelet inhibition
* Smoking
* Blood thinners
* Heart failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Changes in ethanol concentrations before and after omeprazol usage | four weeks
  mM (serum, intestinal fluid, urine and feces)
Changes in fructose concentrations in peripheral blood before and after omeprazol usage | 4 weeks
  Area under the curve of fructose in peripheral blood upon ingestion of 1 gram / kg unlabeled fructose in combination with 1000mg of D-fructose-13C6 measured during fructose challange test
Changes in fructose metabolites in breath before and after omeprazol usage | 4 weeks
  Area under the curve of various metabolites (e.g. ethanol) will be measured in breath samples upon ingestion of 1 gram / kg unlabeled fructose in combination with 1000mg of D-fructose-13C6 measured during fructose challange test
Fructose metabolites in feces before and after omeprazol usage | 4 weeks
  Using 24h feces, the investigators will measure fecal concentrations of fructose metabolites such as ethanol, as well as short chain fatty acids (SCFAs) and bile acids.
Fructose metabolites in urine | 4 weeks
  Using 24h urine, the investigators will measure fecal concentrations of fructose metabolites such as ethanol, as well as SCFAs and bile acids.
Changes in serum glucose concentrations before and after omeprazol | 4 weeks
  mmol/l measured during fructose challange test

SECONDARY OUTCOMES:
Changes in microbiota composition in luminal samples | four weeks
  changes in relative abundance (%) of bacterial phyla, genera and species between groups and after intervention with omeprazol measured by 16sRNA sequencing and shotgun metagenome analysis
Changes in dietary intake | four weeks
  Participants are asked to fill out an online dietary questionnaire for the 3 days prior to study visits
Bioreactor analyses | four weeks
  Using specific anaerobic culturing, ethanol production of fecal samples will be assessed of bacterial strains.
Changes in Oral microbiota composition | four weeks
  changes in relative abundance (%) of bacterial phyla, genera and species between groups and after intervention with omeprazol measured by 16sRNA sequencing.
Differences in gene expression in small intestinal biopsies | 4 weeks
  measured by RNA sequencing
Changes in Fecal microbiota composition | 4 weeks
  changes in relative abundance (%) of bacterial phyla, genera and species between groups and after intervention with omeprazol measured by 16sRNA sequencing and shotgun metagenome analysis
Changes in abundance of post prandial plasma metabolites | 4 weeks
  Postprandial plasma samples will be prepared for the analysis of mainly: organic acids, amino acids, fatty acids, uric acid, glucose and fructose before and after intervention with omeprazol

CONTACTS AND LOCATIONS:
Overall Officials: Max Nieuwdorp, prof, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No